CLINICAL TRIAL: NCT04314362
Title: A Single-center, Vehicle-controlled, Study to Evaluate Methods to Enhance AZR-MD-001 for Meibomian Gland Dysfunction (MGD)
Brief Title: Methods to Enhance AZR-MD-001 for Meibomian Gland Dysfunction (MGD)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Azura Ophthalmics (Industry)
Collaborators: The University of New South Wales (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SOVS2020-080
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Results first posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2020-03

CONDITIONS: Meibomian Gland Dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AZR-MD-001 Active (Experimental): AZR-MD-001 ointment/semi-solid drug (1.0%)
  Interventions: Drug: AZR-MD-001 ointment/semi-solid drug
- AZR-MD-001 Active + Conventional Treatment (Experimental): AZR-MD-001 ointment/semi-solid drug (1.0%) plus Hylo-Forte®
  Interventions: Drug: AZR-MD-001 ointment/semi-solid drug
- AZR-MD-001 vehicle (Experimental): AZR-MD-001 vehicle control
  Interventions: Drug: AZR-MD-001 ointment/semi-solid drug

INTERVENTIONS:
Drug: AZR-MD-001 ointment/semi-solid drug — AZR-MD-001 (1.0%) and suitable excipient

SUMMARY:
Single-center, single-masked (the individual(s) performing efficacy and safety measures will be masked to treatment assignment for the patient(s) they are assessing), vehicle-controlled, randomized study.

DETAILED DESCRIPTION:
Randomized study with 6 visits. For all dose groups a screening visit will be followed by a baseline visit 14 days later (qualification period). At the end of the qualification period patients who still exhibit signs of Meibomian Gland Dysfunction (MGD) at the baseline visit will be enrolled into a 3-month treatment period. At the baseline (Day 0) visit, patients will be randomly assigned to receive either AZR-MD-001 ointment/semi-solid drug or AZR-MD-001 vehicle twice-weekly.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of meibomian gland obstruction (based on a meibomian gland secretion (MGS) score of ≤12 for 15 glands of the lower lid) in both eyes at the baseline visit
* Reported dry eye signs and symptoms within the past 3 months:

Ocular Surface Disease Index (OSDI) score ≥ 13; TBUT < 10 seconds in both eyes

Exclusion Criteria:

* Uncontrolled ocular disease (except for MGD) or uncontrolled systemic disease
* Patient has glaucoma or ocular hypertension as demonstrated by an intraocular pressure (IOP) in either eye at screening of ≥24 mm Hg determined by Goldman applanation tonometry or has planned insertion/removal of glaucoma filtration shunts/devices during the study
* Corneal abnormality or disorder that impacts normal spreading of the tear film (keratoconus, pterygia, scarring) or corneal integrity
* Recent (within the past 3 months of the baseline visit) ocular surgery, trauma, herpes, or recurrent inflammation
* Contact lens use anticipated during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2021-01-06 (Actual); Study Completion 2021-01-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fiona Stapleton, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AZR-MD-001 Active | AZR-MD-001 Vehicle
Started (The results with and without Hylo-Forte were to be combined if Hylo-Forte did not significantly impact safety or efficacy results. The groups were combined for presentation of the results as Hylo-Forte did not significantly impact the observed safety or efficacy results.) | 21 (3 patients were randomized, but did not receive treatment (2 in active 1 in vehicle).) | 11
Completed | 12 | 10
Not Completed | 9 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZR-MD-001 Active | AZR-MD-001 Vehicle | Total
Number analyzed (Participants) | 21 | 11 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (18.9) | 51.2 (16.7) | 47.5 (18.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 6 | 22
  Male | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 6 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 8 | 5 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  Australia | 21 | 11 | 32

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy for MGD: Change From Baseline to Month 3 in Meibomian Gland Secretion Score (MGS)
Description: The MGS can range from 0 (highly abnormal) to 45 (Normal). Meibomian gland assessment was completed using a handheld instrument, Meibomian Gland Evaluator, along the eyelid margin to ensure measurement consistency. A total of 15 glands were evaluated along the lower eyelid margin, consisting of 5 glands located in each of the temporal, central and nasal regions. For each of the 15 glands, expressed secretion characteristics were graded on a 0-3 scale using the published methods from Lane and Colleagues (2012)
  Lane SS, DuBiner HB, Epstein RJ, et al. A new system, the LipiFlow, for the treatment of meibomian gland dysfunction (MGD). Cornea. 2012; 31(4): 396-404.
Time Frame: Month 3
Population: Modified Intent to Treat
Measure: Mean (Standard Deviation); unit: Units on the MGS Scale
Arm/Group | AZR-MD-001 Active | AZR-MD-001 Vehicle
Number analyzed (Participants) | 17 | 10
Units on the MGS Scale | 12.8 (11.3) | 8.8 (5.6)

ADVERSE EVENTS:
Time Frame: 3 Months
Arm/Group | AZR-MD-001 Active | AZR-MD-001 Vehicle
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/10
Other Adverse Events (participants affected / at risk) | 14/19 | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZR-MD-001 Active (N=19) | AZR-MD-001 Vehicle (N=10)
Eye Pain (Eye disorders) | 9 (13) | 1 (2)
Eye Irritation (Eye disorders) | 3 (6) | 1 (1)
Ocular Discomfort (Eye disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/62/NCT04314362/Prot_SAP_000.pdf